CLINICAL TRIAL: NCT06815354
Title: Comprehensive Assessment of Cancer Theranostic Response; Investigating the Intent to Change Treatment Decisions Based on TRAQinform Theranostics
Brief Title: Comprehensive Assessment of Cancer Theranostic Response
Acronym: TRAQinform
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AIQ Solutions (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Weill Medical College of Cornell University (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AIQ 24-3216; 5R44CA285006-02 (NIH)
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Theranostics; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Recruited patients will receive a PSMA PET/CT at week 12 in addition to SOC baseline PSMA PET/CT and diagnostic CT and week 12 diagnostic CT images.
  After each follow-up PET/CT, the local team will make a clinical decision about the care of the patient, using the PET/CT images and other relevant clinical data, but without information provided by TRAQinform Theranostics, and answer a investigator questonnaire. The design is modeled after intent-to-change studies con-ducted by the National Oncology PET Registry (NOPR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Metastatic Prostate Cancer (Other): 32 patients with metastatic prostate cancer planned to start treatment with 177Lu-PSMA (Pluvicto) will be enrolled.
  Interventions: Device: TRAQinform Theranostics

INTERVENTIONS:
Device: TRAQinform Theranostics — This prospective, multi-center, non-interventional clinical study will evaluate actionable outputs from TRAQinform Theranostics, a software only medical device that identifies, quantifies, tracks, and compares lesions between different imaging modalities and multiple imaging timepoints.

SUMMARY:
The intent of this study is to evaluate actionable outputs from TRAQinform Theranostics in a prospective, multi-center, non-interventional clinical study. The primary objective is to investigate intent-to-change treatment decisions after the addition of TRAQinform Theranostics. The exploratory objective is to investigate if treatment efficacy and treatment-related toxicity could be detected by TRAQinform Theranostics following PSMA PET/CT at week 12.

DETAILED DESCRIPTION:
To fully understand the clinical impact of TRAQinform Theranostics on a clinical workflow, this prospective, multi-center, non-interventional clinical study will evaluate actionable outputs from TRAQinform Theranostics, a software only medical device that identifies, quantifies, tracks, and compares lesions between different imaging modalities and multiple imaging timepoints. The primary objective of this clinical study is to investigate intent-to-change treatment decisions after the addition of TRAQinform Theranostics.

The exploratory objective is to investigate if treatment efficacy and treatment-related toxicity can be detected by TRAQinform Theranostics in week 12 of 177Lu-PSMA (Pluvicto) treatment.

This clinical study will enroll 32 metastatic prostate cancer patients, planned to start treatment with 177Lu-PSMA (Pluvicto). Enrolled subjects will receive a 68Ga-PSMA or 18F-DCFPyL PET/CT and a diagnostic CT at baseline (SOC) and again at week 12 of the 177Lu-PSMA treatment. Week 12 PET/CT is for research purposes only and the 68PSMA or 18F-DCFPyL imaging agent may be considered investigational.

Following each imaging timepoint, scans will be transmitted to AIQ for analysis. At baseline and again at week 12, the investigator team, using the PET/CT and other relevant clinical data, will make a treatment decision without TRAQinform Theranostics and complete a questionnaire .

The TRAQinform Theranostics report will then be sent to the investigator team after the patient's treatment decision is made and the team again, will then provide answers to the questionnaire assessing how TRAQinform Theranostics would have impacted treatment decisions.

To address the status quo bias of each local investigator team, a blinded clinical evaluation of the week 12 questionnaire and any other anonymized clinical data necessary to make a treatment decision (prior taxane treatments, relevant labs, physical examination, treatment toxicities, and recent medical history) will be shared with each site. The investigator teams at each site will independently answer the week 12 questionnaire considering all information but without knowledge of the treatment decision made by the investigator teams at the other site.

It is important to note that the objective of this clinical study is to evaluate only the "intent" to change treatment. The investigator teams agree that patient treatment management decisions will not be affected by the additional information from TRAQinform Theranostics, and no clinical intervention will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and willing and able to provide informed consent.
* Diagnosis of metastatic prostate cancer.
* Planned to start 177Lu-PSMA (Pluvicto).
* Ability to tolerate two 68Ga-PSMA or 18F-DCFPyL PET/CT imaging procedures. One at baseline and at 12 weeks of 177Lu-PSMA (Pluvicto) treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 at screening.

Exclusion Criteria:

* Any concurrent disease, infection, or comorbid condition that interferes with the ability of the patient to participate in the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Investigate intent to change treatment decisions after the addition of the TRAQinform Theranostics | 12 weeks
  Medical teams make a treatment decision using the PSMA PET/CT, diagnostic CT, and other clinical data without the TRAQinform Theranostics analysis report. A treatment decision questionnaire is completed. The medical team is then given the TRAQinform Theranostic report, and the treatment decision questionnaire is completed again.
  TRAQinform Theranostic analyzes PSMA PET/CT and CTs. A pdf report allows a medical team to view and interpret the TRAQinform outputs. The report is a theranostic tracer concordance analysis of the PSMA PET/CT and the diagnostic CT for lesions and organs. PSMA PET/CT metrics include SUVmax, SUVmean, Volume and Slice. CT metrics include Volume and Slice. Treatment decisions with/without TRAQinform Theranostics report will be evaluated by calculating the Kappa Index, reported with corresponding 95% confidence interval. Logistic regression analysis will be conducted to correlate decisions with outcomes.

SECONDARY OUTCOMES:
Investigate if treatment efficacy and treatment-related toxicity could be detected by the TRAQinform Theranostics | 12 weeks
  Clinical reports and patient history information from the PRRT patient dataset will be used to identify patients with PRRT-related toxicities (nephrotoxicity, xerostomia, bone pain flair, thrombocytopenia). Toxicity type, grade, and date of first known presence of toxicity will be captured. In addition to identifying single imaging metrics that may predict toxicity, an updated TRAQinform Profile model will be trained to predict patient toxicity status using baseline only imaging and dosimetry metrics and a combination of baseline, follow-up, and response metrics.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Weill Medical College of Cornell, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas